CLINICAL TRIAL: NCT04945876
Title: Effect of Mobile Health Technology (mHealth), Exercise Adherence and Optimal Nutrition Post Rehabilitation Among People With Parkinson's Disease
Brief Title: Exercise Adherence and Optimal Nutrition Post Rehabilitation Among People With Parkinson's Disease
Acronym: mHEXANUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Unicare Fram (Unknown); Norwegian Parkinson's Association (Unknown); Lovisenberg Diaconal University College (Other); Karolinska Institutet (Other); Aalborg University Hospital (Other); Fysiofondet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201660 mHEXANUT
Record Dates: First submitted 2021-03-01; First posted 2021-06-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; digital follow up; exercise; nutrition
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized, controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The complex intervention makes masking of participants and care provider impossible. An independent therapist will conduct baseline testing before randomization. The same therapist will conduct the re-testing at 12 weeks and six month, the assessor will be blinded to group allocation and not be part off providing the intervention. The person conducting the data-analyzes will be blinded to group allocation.
  A computer-generated, permuted block randomization scheme will be used to allocate patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Participants is encouraged to follow the home-based rehabilitation plan based on the recommendations from the rehabilitation center. No further follow up except for testing at 12 weeks and six months.
  After the completion of the study the control group will be offered a session of individual exercise and diet guidance as well as a period of digital follow-up as needed.
- Intervention group (Experimental): Participants will receive a session of individual exercise and diet guidance with focus on goals and motivation for diet and exercise and help to overcome any barriers for self-efficacy. They will also receive an activity tracker and an introduction on how to use it. Further they will receive a monthly digital follow-up to provide support and address questions and goals regarding nutrition, daily energy expenditure and exercise. The participants can also send sms if they have questions during the follow-up period. They will be encouraged to continue to follow the home-based rehabilitation plan based on the recommendations from the rehabilitation center. If needed they can get help to find suitable exercise groups in their own municipality. The Garmin wristband will be used to facilitate daily activity and continuing exercise at recommended intensity level at home. Participants who are malnourished, or at risk of malnutrition, will receive specific guidance session on nutrition.
  Interventions: Behavioral: Digital follow-up

INTERVENTIONS:
Behavioral: Digital follow-up — Participants will receive:
  One session of individual exercise and diet guidance focusing on goals and motivation.
  An activity tracker and instructions on how to use it both for motivation, daily activity tracking, logging of specific exercise and using the wristbands heart rate monitor to control intensity level during exercise.
  Monthly digital follow-up to provide support and address questions and goals regarding nutrition, daily energy expenditure and exercise.
  Opportunity to send sms with questions regarding nutrition and exercise. Participants who are malnourished, or at risk of malnutrition will be offered a total of two hours of additional individualized, digital guidance on nutrition as needed.
  Arms: Intervention group

SUMMARY:
A randomized, controlled trial to evaluate the effect of six months digital follow-up, after a stay at a rehabilitation center, on functional and nutritional status in people with Parkinson Disease.

DETAILED DESCRIPTION:
It is found that regular, structured exercise is especially important for people with Pakinson disease (PD) and it is a key element in the treatment of PD at rehabilitation centers in Norway. A substantial amount of research indicate that exercise can lead to improvements in physical functioning, strength, balance, gait, and HRQOL among people with PD. However, after a supervised exercise period, these measures tend to return toward baseline values. This regression may to some extent reflect the progressive nature of PD, but previous research suggests that maintaining the motivation to stay physically active is difficult once formalized interventions end. Furthermore, research indicate that nutritional status is an important predictor for health status among people with PD and that PD patients have high rates of unintentional weight loss compared to age-matched controls. In other words, research indicate that follow-up at home after rehabilitation is necessary to increase optimal nutrition and continuing to exercise.

This is a randomized controlled trial meant to evaluate the effect of six months digital follow-up, after a 3-5 week stay at a inpatient rehabilitation center, on functional and nutritional status in people with PD.

Eligible participants will be recruited from Unicare Fram Rehabilitation center by a physical therapist and research assistant in collaboration with Unicare Fram employees and a Ph.D student. Informed consent from the participants is obtained from persons with no previous relationship to the patients, and who are not included in their daily treatment, mainly the research assistant. After baseline testing the participants will be randomly allocated to an intervention- or control group.

The intervention in this study is designed to increase the level of adherence after rehabilitation by implementing factors that previous studies have proven successful such as education, goal setting, follow-up from health care personnel and use of mHealth Technology. The intervention consist of 2 phases.

Phase 1: All participants will receive the rehabilitation program currently provided at Unicare Fram rehabilitation center. This is a comprehensive and interdisciplinary rehabilitation program with focus on self-management of the disease including exercise and nutrition.

Phase 2: The control group will receive no further follow-up. The intervention group will receive digital follow up once a month focusing on goals and motivation, and an activity tracker and instructions on how to use it both for motivation, daily activity tracking, logging of specific exercise and intensity control.

All participants will be retested after 12 weeks and 6 months at Unicare Fram rehabilitation center by the research assistant.

Descriptive data will be reported for variables of interest. The data will be analyzed following the intention to treat principle. Prospective differences in primary and secondary outcomes and baseline characteristics between the intervention group and the control group will be assessed by t-tests for continuous and normal distributed variables and with non-parametric tests for categorical variables. Multiple linear and logistic regression modelling will be used to control for confounding of between-group differences. The latest version of Statistical Package of the Social Sciences (SPSS) will be used.

ELIGIBILITY:
Inclusion Criteria:

* >40 years
* Living at home
* Living max 2,5 hours travel distance from Unicare Fram
* A diagnosis of idipathic PD
* Hoehn-Yahr stage 1-3
* eternal feeding ability
* must own a smart phone

Exclusion Criteria:

* Hoehn-Yahr stage 4-5
* Medical issues that might affect participation in exercise programs
* Diagnosis of dementia
* Diagnosis of severe dysphagia
* Exercises regularly more than twice a week(structured exercise).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Six minute walk test (6MWT) | measured at baseline, 12 weeks and 6 months
  A sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. It evaluates the functional capacity of the individual.

SECONDARY OUTCOMES:
The Parkinson's disease questionnaire (PDQ-39) | measured at baseline, 12 weeks and 6 months
  A 39 item, patient reported measure of health status and quality of life over the last month. It assesses how often people affected by parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. The answers results in a score from 0-100 points in each dimension. Lower scores reflect better QoL.
The Patients-Generated subjective Global Assessment Short Form (PG-SGA) | measured at baseline, 12 weeks and 6 months
  It is a component of a nutritional assessment tool wich could be used for descriptive nutrition screening. A 4 item questionnaire assessing weight, food-intake, symptoms affecting food intake and activity & function. The answers result in a score from 0-9, 0 indicates no need for nutritional measures, 9 indicates a critical need for nutritional measures.
mini best test | measured at baseline, 12 weeks and 6 months
  The test is used to identify risk of falling, changes in balance over time and distinguish between different balance challenges.
and 5x sit-to-stand | measured at baseline, 12 weeks and 6 months
  Assesses functional lower extremity strength, transitional movements, balance and fall risk
Bioelectrical impedance analysis | measured at baseline, 12 weeks and 6 months
  A method for estimating body composition, in particular body fat and muscle mass.
What do you eat | measured at baseline
  A food frequency questionnaire used to assess the diet of a population during the last seven days. Contains questions on how often and how much you eat of specific food groups. The questionnaire does not result in a score. it can be used to raise awareness and to assess on what areas potential nutritional measures is needed.
Radboud Oral Motor Inventory for Parkinson's disease (ROMP) - swallowing | measured at baseline, 12 weeks and 6 months
  A self-report questionnaire with 7 questions assessing potential swallowing difficulties. The answers results in a score from 7-35 point. A low score indicates little to no problems with swallowing, i high score indicates a higher degree of problems with swallowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Unicare Fram Rykkin, Rykkin, Bærum, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alnes SR, Laerum-Onsager E, Bye A, Vistven A, Franzen E, Holst M, Brovold T. Mobile health technology, exercise adherence and optimal nutrition post rehabilitation among people with Parkinson's Disease (mHEXANUT) - a randomized controlled trial protocol. BMC Neurol. 2023 Mar 2;23(1):93. doi: 10.1186/s12883-023-03134-5. PMID 36864377